CLINICAL TRIAL: NCT02217267
Title: Long Term Outcome After Serial Lidocaine Infusion in Peripheral Neuropathic Pain : A Pilot Study
Brief Title: Long Term Outcome After Serial Lidocaine Infusion in Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI140/2014
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Neuropathy
Keywords: Peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Normal Saline 50 ml intravenous infusion in 1 hour once a week 4 times
  Interventions: Drug: Placebo
- Lidocaine group (Active Comparator): Lidocaine 3mg/kg in Normal Saline to 50 ml intravenous infusion in 1 hour once a week 4 times
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 3 mg/kg dilute in Normal Saline to 50 ml intravenous infusion in 1 hour
  Other Names: Intravenous lidocaine
  Arms: Lidocaine group
Drug: Placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study to evaluated Long term outcome after serial Lidocaine infusion when compared with placebo in peripheral neuropathic pain patients in acute stage (less than 6 months) at 3 months after first time of infusion

DETAILED DESCRIPTION:
Peripheral nerve injury may give rise to severe and long-lasting types of pains which are often resistant to treatment such as opioid, tricyclic antidepressant or anticonvulsant. Lidocaine infusion has been the one of intractable neuropathic pain treatment . My hypothesis the serial lidocaine infusion can adequate pain control and can prevent chronic pain (central sensitisation). Therefore, we designed this prospective, randomised, double-blind, controlled study to evaluate the efficacy of serial lidocaine infusion in peripheral neuropathic pain compared with placebo in long term outcome (at 3 month).

ELIGIBILITY:
Inclusion Criteria:

* Peripheral neuropathic pain from peripheral nerve injury within 6 months after injury
* Well understand to Thai language in writing or listening

Exclusion Criteria:

* Underlying Heart disease or Arrhythmia
* Allergy to lidocaine, Gabapentin, Carbamazepine, tramadol
* History of epilepsy
* History of lidocaine used
* Underlying Psychiatric disease
* History of drug abuse
* Pregnancy and nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08-01; Primary Completion 2017-12-29 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity | at 3 months after serial lidocaine infusion
  Pain intensity (Numerical Rating Scale; from 0-10) 0 means no pain, and 10 means worst pain imaginable.

SECONDARY OUTCOMES:
Quality of life using Utility score | at 3 month after serial lidocaine infusion
  Quality of life will be assessed using EuroQol5D5L and reported as a utility score (0-1.0) "0" represents death, and "0.1" means full health

OTHER OUTCOMES:
Psychological effects on depression, anxiety and stress | at 3 month after serial lidocaine infusion
  The psychological effect will be assessed using DASS21. Each of these domains is assessed with a separate 7-item scale. Responses to the items are summed to create scales with a total possible score of 21 points, then multiplied by two to calculate the final score. The final score can then be graded in each domain: Normal (0-4), Mild (5-6), Moderate (7-11), Severe (11-13), and Extremely Severe (14+) for depression; Normal (0-3), Mild (4-5), Moderate (6-7), Severe (8-9) and Extremely Severe (10+) for anxiety; and Normal (0-7), Mild (8-9), Moderate (10-12), Severe (13-16) and Extremely Severe (14+) for stress.

CONTACTS AND LOCATIONS:
Overall Officials: Suratsawadee Wangnamthip, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Result] Challapalli V, Tremont-Lukats IW, McNicol ED, Lau J, Carr DB. Systemic administration of local anesthetic agents to relieve neuropathic pain. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD003345. doi: 10.1002/14651858.CD003345.pub2. PMID 16235318
- [Result] Attal N, Rouaud J, Brasseur L, Chauvin M, Bouhassira D. Systemic lidocaine in pain due to peripheral nerve injury and predictors of response. Neurology. 2004 Jan 27;62(2):218-25. doi: 10.1212/01.wnl.0000103237.62009.77. PMID 14745057
- [Result] Kingery WS. A critical review of controlled clinical trials for peripheral neuropathic pain and complex regional pain syndromes. Pain. 1997 Nov;73(2):123-139. doi: 10.1016/S0304-3959(97)00049-3. PMID 9415498
- [Result] Wallace MS, Dyck BJ, Rossi SS, Yaksh TL. Computer-controlled lidocaine infusion for the evaluation of neuropathic pain after peripheral nerve injury. Pain. 1996 Jul;66(1):69-77. doi: 10.1016/0304-3959(96)02980-6. PMID 8857633
- See also: Siriraj Institutional Review Board — http://www.si.mahidol.ac.th/th/division/sirb/